CLINICAL TRIAL: NCT03853915
Title: FDG-PET and Circulating HPV in Patients With Cervical Cancer Treated With Definitive Chemoradiation (II)
Acronym: HPVDNA02
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-6277
Record Dates: First submitted 2019-02-22; First posted 2019-02-26 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; PET Scan; HPV DNA
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Newly diagnosed FIGO stage IB-IVA cervical cancer patients planned for definitive chemoradiation will be accrued to study and will have:
  1. FDG PET Scan at 3 month time point.
  2. Blood sample to measure HPV DNA at time point baseline, end of radiotherapy, 4-6 weeks and 3 months post completion of definitive radiotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FDG PET Scan (Experimental): [F-18] - FDG PET Scan and blood sample to measure HPV DNA
  Interventions: Diagnostic Test: [18-F]- FDG - PET

INTERVENTIONS:
Diagnostic Test: [18-F]- FDG - PET — [F-18]-FDG Injection is an intravenous diagnostic radiopharmaceutical used for Positron Emission Tomography. While this is not the subject of investigation in this study, [F-18]-FDG will be used in the PET imaging assessment of study participants during their 3 month follow-up post-treatment.

SUMMARY:
Nearly all cervical cancers are caused by the human papilloma virus (HPV), which can be detected in cancer tissue by laboratory tests. There is evidence that the virus can also be detected from a blood sample to monitor the effects of treatment. Previous studies have shown that a special test called 18F-Fluorodeoxyglucose (FDG) Positron Emission Tomography/Computed Tomography (PET-CT) at 3 months after treatment may predict survival in cervical cancer.

The purpose of this study is to see how well the FDG-PET Scan and blood tests for HPV can detect leftover cervical cancer cells after treatment. This study is not a particular form of treatment and patients will receive standard of care treatment.

DETAILED DESCRIPTION:
Cervical cancer is the 4th most common malignancy in women worldwide. A significant proportion of women with locally advanced cervical cancer are primarily managed with chemotherapy and radiotherapy which has improved the 5-year survival and disease-free survival; however both local and distant recurrences still remain to be challenges after treatment.

A prospective study has shown that metabolic response on post-therapy FDG-PET scan at 3 months to be predictive of progression-free and overall survival in patients with locally advanced cervical cancer. It may also predict patterns of failures for these patients.

HPV is recognized as a necessary cause of the vast majority of cervical cancer and HPV DNA has been detected in circulation from patients with cervical cancer and oropharyngeal cancer at diagnosis and at the time of relapse. Despite the promising potential of HPV DNA to monitor response and detect recurrence at an early stage, no study has evaluated serial HPV DNA and its association with PET response and survival.

We have recently reported preliminary data from a feasibility study (HPVDNA01) on 20 patients. Detectable HPV DNA at the end of cervical radiation therapy predated the clinical diagnosis of metastases and was associated with inferior progression-free survival. Also, 3 month plasma HPV DNA level was more accurate than 3-month FDG PET imaging in detecting leftover disease. This follow-up study aims to validate the clinical utility of plasma HPV DNA detection.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma of the cervix, FIGO stage IB-IVA
* 3.1.2 Planned for radical radiotherapy and concurrent cisplatin chemotherapy.
* 3.1.3 Age ≥ 18 years.

Exclusion Criteria:

* Evidence of distant metastases (suspicious paraaortic nodes below the renal vessels allowed if they will be encompassed within the radiation field)
* Patients who have received any anticancer treatment for their cervical cancer.
* Other cervical cancer tumor histologies (e.g. small cell, serous)
* Contraindications to 18FDG PET-CT
* Contraindication to radiotherapy (e.g. severe Crohn's disease)
* Contraindication to chemotherapy (e.g. non-reversible renal failure)
* History of another invasive malignancy, except for non-melanoma skin cancer or tumors curatively treated with no evidence of disease for ≥ 5 years.
* Known pregnancy or lactating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-04-23 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate | up to 5 years
  The progression-free survival rate of patients with and without detectable plasma HPV DNA post treatment

SECONDARY OUTCOMES:
Plasma HPV DNA levels | Up to 3 months
  The accuracy of 3-month FDG-PET or 3-month HPV DNA for predicting relapse will be estimated.

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, The Princess Margaret, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han K, Zou J, Zhao Z, Baskurt Z, Zheng Y, Barnes E, Croke J, Ferguson SE, Fyles A, Gien L, Gladwish A, Lecavalier-Barsoum M, Lheureux S, Lukovic J, Mackay H, Marchand EL, Metser U, Milosevic M, Taggar AS, Bratman SV, Leung E. Clinical Validation of Human Papilloma Virus Circulating Tumor DNA for Early Detection of Residual Disease After Chemoradiation in Cervical Cancer. J Clin Oncol. 2024 Feb 1;42(4):431-440. doi: 10.1200/JCO.23.00954. Epub 2023 Nov 16. PMID 37972346